CLINICAL TRIAL: NCT07215845
Title: Pars Healing on oZTEo MRI
Brief Title: Pars Healing on MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Lauren Pringle, Assistant Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2127781
Record Dates: First submitted 2025-09-16; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pars Interarticularis Stress Fracture; Pars Interarticularis Stress Injury
Keywords: MRI; Pars Interarticularis Stress Fracture; Pars Interarticularis Stress Injury; Pars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Group (Experimental): Participants will receive serial MRIs over the course of 12-months at 2-, 4-, 6-, and 12 month intervals. This group's images will be used to help guide their clinical care outcomes.
  Interventions: Device: MRI
- Control Group (Other): Participants will receive serial MRIs over the course of 12-months at 2-, 4-, 6-, and 12 month intervals. This group's images will NOT be used to help guide their clinical care outcomes for the 2-, 4-, and 6-month images. However, the 12-month images may be used to guide clinical care outcomes.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Reader confidence using standard lumbar MRI techniques on diagnosing pars stress injuries will be compared to advanced techniques. Additionally, various software/MRI sequences will be tested to evaluate image quality and to improve resolution compared to institution pars MRI scan protocols.

SUMMARY:
The goal of this clinical trial is to learn more about the natural healing process of pars stress injuries in adolescents and young adults by documenting bony bridging across stress fractures using Magnetic Resonance Imaging (MRI). It is hypothesized that many of these injuries can and will heal with appropriate rest and rehabilitation. Long-term, it is hoped that follow-up MRI exams can help guide clinical management by visualizing the healing and allowing individuals to return to play after bony bridging has occurred.

Participants will be asked to undergo serial MRI scans over the course of a 12-month period and answer a brief questionnaire at each visit.

DETAILED DESCRIPTION:
There is not a current, well-established standard of care (SoC) for initial diagnosis or follow-up imaging worldwide and these injuries are likely underdiagnosed. Some practices use conventional Magnetic Resonance Imaging (MRI) sequences which can be challenging to interpret, and the patient may undergo repeat testing or alternative imaging including Computed Tomography (CT), bone scans, or repeat MRIs (the former two of which can be high radiation and not optimal at the young age group).

ELIGIBILITY:
Inclusion Criteria:

* 12-30 years old
* Symptoms of back pain at the time of enrollment
* Clinical imaging demonstrating pars stress interarticularis injury or pars interarticularis defect

Exclusion Criteria:

* Prior lumbar surgery
* Any condition for which an MRI procedure is contraindicated (e.g., metallic material in the body such as pacemakers, metallic clips, etc.)
* Pregnancy
* Likelihood of claustrophobia
* Any patient-related factors that compromised quality on the initial diagnostic scan (patient motion, ascites fluid, difficulty with positioning during the scan)

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pars Stress Injury Healing | From enrollment to 12 months (4 total research scans at 2 months, 4 months, 6 months, and 12 months post initial scan)
  Stress injuries (fracture line and/or bone marrow edema) identified prior to study enrollment via initial clinical MRIs will be followed over serial research MRIs at 2 months, 4 months, 6 months, and 12 months after initial clinical MRI was completed. At each MRI, the fracture morphology (incomplete vs complete), bony bridging across any fracture line previously seen, amount of sclerosis, and presence of bone marrow edema will be described to assess degree of injury healing. Patient questionnaires including questions on pain scores will also be administered at the time of the research MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Pringle, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
By signing the consent form, participants will be providing consent to the study team for their information to be shared with other researchers without obtaining their consent again. If/when data is shared with other researchers outside of the study, individual participant data will be de-identified as to not share the identity of participants. The IDP to be shared would be participant's MRI images and answers to study questionnaires.

REFERENCES:
- [Background] Aydingoz U, Yildiz AE, Ergen FB. Zero Echo Time Musculoskeletal MRI: Technique, Optimization, Applications, and Pitfalls. Radiographics. 2022 Sep-Oct;42(5):1398-1414. doi: 10.1148/rg.220029. Epub 2022 Jul 29. PMID 35904982
- [Background] Watura C, Mitchell AWM, Fahy D, Houghton J, Kang S, Lee JC. T1-VIBE and STIR MRI of lumbar pars interarticularis injuries in elite athletes: fracture characterisation and potential prognostic indicators. Skeletal Radiol. 2024 Mar;53(3):489-497. doi: 10.1007/s00256-023-04437-x. Epub 2023 Aug 31. PMID 37650925
- [Background] Ang EC, Robertson AF, Malara FA, O'Shea T, Roebert JK, Schneider ME, Rotstein AH. Diagnostic accuracy of 3-T magnetic resonance imaging with 3D T1 VIBE versus computer tomography in pars stress fracture of the lumbar spine. Skeletal Radiol. 2016 Nov;45(11):1533-40. doi: 10.1007/s00256-016-2475-7. Epub 2016 Sep 10. PMID 27614965
- [Background] Schwaiger BJ, Schneider C, Kronthaler S, Gassert FT, Bohm C, Pfeiffer D, Baum T, Kirschke JS, Karampinos DC, Makowski MR, Woertler K, Wurm M, Gersing AS. CT-like images based on T1 spoiled gradient-echo and ultra-short echo time MRI sequences for the assessment of vertebral fractures and degenerative bone changes of the spine. Eur Radiol. 2021 Jul;31(7):4680-4689. doi: 10.1007/s00330-020-07597-9. Epub 2021 Jan 14. PMID 33443599
- [Background] Standaert CJ. Spondylolysis in the adolescent athlete. Clin J Sport Med. 2002 Mar;12(2):119-22. doi: 10.1097/00042752-200203000-00009. No abstract available. PMID 11953559
- [Background] Vij N, Naron I, Tolson H, Rezayev A, Kaye AD, Viswanath O, Urits I. Back pain in adolescent athletes: a narrative review. Orthop Rev (Pavia). 2022 Aug 5;14(3):37097. doi: 10.52965/001c.37097. eCollection 2022. PMID 35936806
- [Background] Murphy KP, Sanders C, Rabatin AE. Evaluation and Treatment of the Child with Acute Back Pain. Pediatr Clin North Am. 2023 Jun;70(3):545-574. doi: 10.1016/j.pcl.2023.01.013. Epub 2023 Mar 21. PMID 37121642